CLINICAL TRIAL: NCT04264715
Title: Evaluation of the Impact of Germicidal Light (Indigo-Clean) on Intraoperative S. Aureus Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Andrew Gostine, MD, Anesthesiologist and Intensivist, Northwestern Medicine
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 19-044
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pathogen Transmission
MeSH Terms: interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 405nm light room (Experimental): In this room, surgeries will be performed under ambient light including the wavelength 405nm
  Interventions: Device: 405nm light
- Control room (No Intervention): In this room, surgeries will be performed under ambient light from regular phosphorescent light does not include 405nm frequencies

INTERVENTIONS:
Device: 405nm light — In this room, surgeries will be performed under ambient light including the wavelength 405nm
  Arms: 405nm light room

SUMMARY:
Operating room S. aureus exposure has been directly linked to postoperative infections and is therefore an important target for infection prevention. Visible light (non-ultraviolet spectrum) at 405nm has been shown to be germicidal. We hypothesize that use of this light in operating rooms will reduce S. aureus transmission occurring within and between patients and reduce surgical site infections (SSIs). Visible light is safe for routine, continual exposure, and is less harmful than sunlight. We plan to install ambient, germicidal lighting in 4 operating rooms. This ambient light is not directly applied to patients (does not involve the surgical procedure lights). Patients will undergo surgery according to usual practice. We will conduct a case-control study where operating rooms with surgeries with the lights are matched to operating rooms with surgeries without lights.

In Aim 1, 4 OR-pairs will be observed each day over an anticipated 103 working days for the primary outcome of S. aureus transmission events over a total minimum study period of 5.2 months (103 working days).

ELIGIBILITY:
Inclusion Criteria:

* Operating Rooms with and without the bactericidal lights where adult patients undergoing orthopedic, cardiothoracic, gynecology/oncology, and neurological surgery.

Exclusion Criteria:

* Operating Rooms with and without the bactericidal lights where pediatric, incarcerated, and/or pregnant patients undergoing surgery outside of the classifications above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 824 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Staphylococcus aureus transmission rate | sequential surgeries on the same 1 day
  We will be assessing the transmission of bacteria to the patient during the case and from previous cases to subsequent cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Lake Forest Hospital, Lake Forest, Illinois, United States

IPD SHARING:
Plan to Share IPD: No